CLINICAL TRIAL: NCT06209645
Title: Non-invasive Analgesic Stimulation of the Patient's Motor Cortex With an Oscillating Electric Current at the Dominant Frequency Recorded by EEG
Brief Title: Non-invasive Personalized Transcranial Cortical Neurostimulation for Pain Relief
Acronym: PERSOSTIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 69HCL23_0810
Record Dates: First submitted 2023-12-06; First posted 2024-01-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-01

CONDITIONS: Drug-resistant Neuropathic Pain
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The study involves the use of transcranial electrical stimulation applied to the motor cortex at each subject's own cortical rhythm. The rhythm is previously obtained by electroencephalographic (EEG) recording. Fifty adult patients, recruited by the Pain Evaluation and Treatment Center of the Neurological hospital, at the Hospices Civils de Lyon, suffering from drug-resistant neuropathic pain for more than 12 months.
  The stimulation (tACS) will be compared head-to-head with another reference active stimulation modality, namely anodal direct current stimulation (tDCS) of the motor cortex. The 2 types of active stimulation will be performed in cross-over mode, in randomized order, and compared with placebo stimulation.
  Each stimulation modality will comprise 6 sessions spaced 2 weeks apart, with the first session in placebo mode and the next 5 in active mode.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS then tACS (Experimental): This group is made up of adult patients with drug-resistant neuropathic pain, who started with tDCS stimulation, followed by tACS stimulation, in accordance with randomization. Each series of each modality comprises 6 sessions spaced 2 weeks apart, the first session being in placebo mode and the following 5 in active mode. Each session lasts 20 minutes. In placebo mode, a 2 miliampere (mA) current is delivered for 30 seconds at the start and at the end of the session, to prevent the patient noticing the difference between placebo and active stimulation. In active mode, the 2mA current is delivered for the duration of the session.
  Interventions: Device: tDCS (Transcranial Direct Current Stimulation); Device: tACS (Transcranial Alternating Current Stimulation)
- tACS then tDCS (Experimental): This group is made up of adult patients with drug-resistant neuropathic pain, who started with tACS stimulation, followed by tDCS stimulation, in accordance with randomization. Each series of each modality comprises 6 sessions spaced 2 weeks apart, the first session being in placebo mode and the following 5 in active mode. Each session lasts 20 minutes. In placebo mode, a 2mA current is delivered for 30 seconds at the start and at the end of the session, to prevent the patient noticing the difference between placebo and active stimulation. In active mode, the 2mA current is delivered for the duration of the session.
  Interventions: Device: tDCS (Transcranial Direct Current Stimulation); Device: tACS (Transcranial Alternating Current Stimulation)

INTERVENTIONS:
Device: tDCS (Transcranial Direct Current Stimulation) — The tDCS group will be treated with non-invasive motor cortex stimulation. A two-minute EEG recording will be made before each session, using the same electrodes as for stimulation. Anodal stimulation of 2,0 mA will be delivered over the motor area contralateral to the painful region (C4 or C3 according to the international 10-20 system). The return electrode will be placed over the fronto-polar region (FP1 or FP2) ipsilateral to the painful region. If pain is bilateral, the most painful region will be chosen to be treated.
Device: tACS (Transcranial Alternating Current Stimulation) — The tACS group will be treated with non-invasive motor cortex stimulation. The stimulation series comprises six sessions spaced 2 weeks apart, the first session being placebo. A two-minute EEG recording will be made before each session, using the same electrodes as for stimulation. Stimulation frequency will be set according to the dominant frequency recorded over the motor area. Anodal stimulation of 2,0 mA will be delivered over the motor area contralateral to the painful region (C4 or C3 according to the international 10-20 system). The return electrode will be placed over the fronto-polar region (FP1 or FP2) ipsilateral to the painful region.

SUMMARY:
Neuropathic pain is a public health problem with less than 50% of patients being relieved by drug treatments.

Surgically implanted motor cortex stimulation represents an invasive therapeutic solution capable of relieving a significant proportion of drug-resistant patients (1 in 2); it cannot, however, be offered to all patients, and is not morbidity-free.

Non-invasive motor cortex stimulation techniques have been refined over the last decade, in particular transcranial repetitive magnetic stimulation (rTMS) and transcranial direct current stimulation (tDCS), which provide pain relief among almost half of drug-resistant patients with few or no side effects.

To be efficient, cortical stimulation requires the activation of multiple distant networks involved in the cognitive and motivational response to pain; stimulation frequency is a crucial parameter for activating these mechanisms. The match between cortical stimulation frequency and the intrinsic neuronal frequency of the stimulated cortex has recently been suggested as a key determinant of clinical effect. Indeed, the transmission efficiency of an oscillatory network increases when its intrinsic frequency matches that of the stimulus applied to it. Given that human sensorimotor networks spontaneously oscillate at frequencies around 10 and 20 Hertz (Hz), this match could underlie the superior efficacy of transcranial stimulation at these frequencies.

The hypothesis of the study is that the analgesic effect of cortical stimulation will be enhanced if the stimulation frequency resonates with the spontaneous oscillations of the underlying cortex, thus facilitating its connectivity with the remote structures involved in pain control. The investigators propose to test this hypothesis in a population of patients with drug-resistant neuropathic pain, referred to the Pain Evaluation and Treatment Center (CETD) of the Neurological hospital, at the Hospices Civils de Lyon. The overall aim of the project is to compare the efficacy of stimulation at each individual's own rate of oscillation of the motor cortex, against a "classic" stimulation protocol, and against placebo stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years
* Neuropathic pain of more than one year's duration1
* Failed treatment with tricyclic or tetracyclic antidepressants, antiepileptics and a combination of morphine and a serotonin (5HT) norepinephrine (NA2) reuptake inhibitor, in the absence of contraindication.
* Average pain intensity of at least 4/10 in the month preceding the inclusion visit.
* Recipient or beneficiary of a social security scheme-

Exclusion Criteria:

* Chronic non-neuropathic pain or pain associated with progressive pathology, active epilepsy, unhealed scalp wound, impaired comprehension or communication that prevents subjective daily and weekly assessments.
* Active epilepsy, treated or not
* Unhealed scalp wound adjacent to EEG recording electrodes or transcranial stimulation application (contraindication to Medical Device (DM) use)
* Pregnant or breast-feeding women
* Inability to understand or follow the ins and outs of the study, in particular the need to assess pain intensity on a daily basis or to trace it, possibly with the help of a third party (comprehension or communication disorders).
* People under guardianship, curatorship or legal protection
* Persons deprived of their liberty, persons under psychiatric care and persons admitted to a health or social establishment for purposes other than clinical investigation
* Participation in other research interfering with the present study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity measure | daily from the beginning until the end of the protocol (15 months)
  Comparison of weekly standardized averages of the Numerical rating scale (NRS) values at the end of tACS versus tDCS versus placebo stimulation sessions.
  Pain scale measurement:
  pain scale : 1 the minimum and 10 maximum value, 10 the higher score mean a worse outcome.

SECONDARY OUTCOMES:
Percentage of responding patients Percentage of patients responding favorably to stimulation (Z-score <-2) after tACS and conventional tDCS. | daily from the beginning until the end of the protocol (15 months)
  The response is considered favorable if on the NRS scale, compared with the baseline of each participant, there is a pain improvement of:
  * more than 30% or
  * more than 2 points or
  * more than 2 Standard Deviation
  Pain scale measurement:
  pain scale : 1 the minimum and 10 maximum value, 10 the higher score means a worse outcome.
Patient's Global Impression of Change (PGIC) Comparison of weekly standardized values of the PGIC at the end of tACS versus tDCS versus placebo stimulation sessions. | one a week from the beginning until the end of the protocol (15 months)
  The PGIC is a seven-points scale that allows the patient to rate their overall impression of change
  1 minimum value and 7 maximum value, and 7 higher score means worse result.
Fatigue score Comparison of weekly standardized averages of the fatigue score values at the end of tACS versus tDCS versus placebo stimulation sessions. | daily from the beginning until the end of the protocol (15 months)
  The fatigue score is a ten-points (from 0 to 10) scale that allows the patient to rate their fatigue
  fatigue scale : 1 the minimum and 10 maximum value, 10 the higher score means a worse outcome.
Sleep score Comparison of weekly standardized averages of the sleep score values at the end of tACS versus tDCS versus placebo stimulation sessions. | daily from the beginning until the end of the protocol (15 months)
  The sleep score is a ten-points (from 0 to 10) scale that allows the patient to rate their quality of sleep with 0= bad quality and 10 = excellent quality
  Sleep scale : 1 the minimum and 10 maximum value, 10 the higher score means a worse outcome.
Sympathetic Skin Response (SSR) measurement Variation, in patients with hyperalgesia/allodynia, of Sympathetic Skin Response after treatment with tACS versus tDCS versus placebo. | SSR will be measured in allodynic patients before each stimulation and evaluation session, starting with the first stimulation session until the end of the protocol (15 months)
  SSR is an objective measure of patient's arousal. For patients suffering from allodynia, SSR will be measured after touch (brush) and/or heat (laser) stimulation on sensitized region and a symmetrical non-sensitised region
  SSR is expressed in mV(millivolt). It is a record of a physiological measurement. The minimum value corresponds to the absence of a response greater than the background recorded by the electrodes. There is no maximum value. The change in response is significant if there is a change greater than 30% from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Charbel SALAMEH, MD, Principal Investigator — Central Integration of pain lab (NeuroPain); Lyon Neurocience research center